CLINICAL TRIAL: NCT07104643
Title: A Phase Ib/II Clinical Study to Evaluate the Safety and Efficacy of TYK-00540 Combined With Enzalutamide in the Treatment of Metastatic Castration-resistant Prostate Cancer (mCRPC) That Has Failed Previous Novel Endocrine Therapy
Brief Title: Study of TYK-00540 Combined With Enzalutamide in Patients With Metastatic Castration-resistant Prostate Cancer（mCRPC）
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYKM5807201
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: mCRPC
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TYK-00540+Enzalutamide (Experimental): Find the maximum tolerated dose(MTD) and the recommended phase 2 dose (RP2D) of TYK-00540, given orally. • Increased dose cohorts from low dose to MTD, starting at 20mg twice a day. Enzalutamide, 160mg each time, once a day.
  Interventions: Drug: TYK-00540; Drug: Enzalutamide

INTERVENTIONS:
Drug: TYK-00540 — Take the specified dose (20mg or 30mg) orally twice a day. Take it on an empty stomach in the morning with about 200 mL of warm water.
Drug: Enzalutamide — Take orally, 160mg each time, once a day. Take orally with or without meals.

SUMMARY:
This study is to evaluate the safety, and preliminary antitumor activity of TYK-00540 combined with Enzalutamide in patients with metastatic castration-resistant prostate cancer (mCRPC) that have failed novel endocrine therapy

DETAILED DESCRIPTION:
This is an open-label, multi-center, dose-escalation and expansion phase Ib/II study to evaluate dose limiting toxicities (DLT) and determine the maximum tolerated dose (MTD) in subjects with metastatic castration-resistant prostate cancer (mCRPC).

To evaluate the efficacy of TYK-00540 combined with Enzalutamide in subjects with metastatic castration-resistant prostate cancer (mCRPC) that have failed novel endocrine therapy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Metastatic castration-resistant prostate adenocarcinoma confirmed by pathology (with no neuroendocrine or small cell features indicated by the initial pathological examination), if pathological examination is performed in the subsequent CRPC stage, the accompanying other pathological types should not exceed 10%. Those with only pelvic lymph node metastasis or local recurrence and metastasis (such as in the bladder, rectum, etc.) cannot be included.
3. At the time of screening, testosterone levels were at castration levels (≤50ng/dL or 1.70nmol/L). If the patient had not previously undergone bilateral orchiectomy, they must be undergoing and voluntarily continue to receive LHRH agonists/antagonists for androgen deprivation therapy throughout the study treatment period.
4. During screening, if the disease progresses, that is, the subject experiences one or more of the following three conditions; PSA progression is defined as no PSA > 1ng/ml and at least two elevated PSA levels with an interval of ≥1 week. ② Disease progression as defined in RECIST 1.1; ③ Bone disease progression as defined by the PCWG3 standard refers to the discovery of ≥2 new lesions on bone scans.
5. Previous anti-tumor treatment must meet the following requirements: having failed in only one approved and marketed novel endocrine therapy in the past (referring to disease progression during the process of novel endocrine therapy; The definition of disease progression is the same as that in inclusion criterion 4), such as abiraterone acetate, apatamide, darotamide or rivelutamide, etc., and no treatment with enzalutamide has been received.
6. ECOG score ≤1, no deterioration in the two weeks prior to study enrollment, and an expected survival period of ≥3 months
7. Have good organ functions, including:

   1. Liver function Total bilirubin (TBIL) ≤ 1.5×ULN (except for documented Gilbert syndrome), alanine aminotransferase (ALT) ≤ 2.5×ULN, and aspartate aminotransferase (AST) ≤ 2.5×ULN (for patients with liver metastasis, ALT/AST≤5×ULN), albumin ≥3.0g/L;
   2. Renal function enhancement: Serum creatinine (Cr) ≤ 1.5×ULN, or creatinine clearance rate ≥50 mL/min;
   3. <S:1> Blood routine: PLT ≥ 100×109/L, ANC ≥ 1.5×109/L, WBC≥ 3.5×109/L and Hb ≥ 90g/L;
   4. The international normalized ratio (INR) is ≤1.5, and the activated partial prothrombin time (APTT) is ≤1.5×ULN;
8. The patient agrees to maintain abstinence (control heterosexual sexual intercourse) or take contraceptive measures, and agrees not to donate sperm;
9. Understand and voluntarily sign the written ICF, and have the willingness and ability to complete regular visits, treatment plans, laboratory tests and other experimental processes.

Exclusion Criteria:

1. Subjects with the following treatments:

   1. Those who have previously received selective CDK2, CDK4 inhibitors, CDK4/6 inhibitors (e.g., Palbociclib, Ribociclib, Abemaciclib, Trilaciclib/G1T38, SHR6390, pirociclib) for treatment;
   2. Previously received enzalutamide or two or more novel endocrine therapies for prostate cancer;
   3. Isotope therapy with strontium-89, samarium or radium-223 was received within 12 weeks prior to the first administration;
   4. Systemic treatment for prostate cancer (anti-androgen therapy, chemotherapy, targeted therapy, immunotherapy, or other interventional clinical trial drugs, except castration therapy drugs) has been received within 4 weeks prior to the first medication.
   5. Systemic treatment for prostate cancer (anti-androgen therapy, chemotherapy, targeted therapy, immunotherapy, or other interventional clinical trial drugs, except castration therapy drugs) has been received within 4 weeks prior to the first medication.
   6. The patient has received blood transfusion, albumin infusion or used hematopoietic growth factor within 2 weeks before the first administration;
   7. Major surgery was performed within 28 days before the first administration of the drug , or surgery was performed when the surgical effect had not yet recovered at the time of screening or during the planned enrollment for treatment;
   8. Has received allogeneic transplants such as stem cell transplantation, bone marrow transplantation or liver transplantation in the past;
   9. Palliative radiotherapy was received within 2 weeks before the first administration;
   10. The first administration was within no more than five half-lives from the implantation of radioactive particles;
   11. The first administration was within no more than five half-lives from the implantation of radioactive particles.
2. In addition to prostate cancer, there are other malignant tumors at the same time (excluding basal cell carcinoma or squamous cell carcinoma of the skin that can be treated locally and have been cured, superficial bladder cancer, cervical carcinoma in situ, ductal carcinoma of the breast and papillary thyroid carcinoma, etc.); Excluding those with other malignant tumors who have been cured of radical treatment for ≥5 years;
3. In addition to prostate cancer, there are other malignant tumors at the same time (excluding basal cell carcinoma or squamous cell carcinoma of the skin that can be treated locally and have been cured, superficial bladder cancer, cervical carcinoma in situ, ductal carcinoma of the breast and papillary thyroid carcinoma, etc.); Excluding those with other malignant tumors who have been cured of radical treatment for ≥5 years;
4. Known to be allergic to any excipients of TYK-00540 tablets, or allergic to enzalutamide and its excipients;
5. Patients whose progression of bone and soft tissue lesions cannot be evaluated, that is, those who simultaneously meet the following two criteria:

   1. The bone scan shows a super bone imaging.
   2. According to RECIST1.1 criteria, there are no assessable soft tissue lesions (measurable or unmeasurable).
6. The patient has any unstable or other disease or medical condition that may affect its safety or compliance with the study, any serious or uncontrolled systemic disease, including uncontrolled hypertension (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥95 mmHg), uncontrolled diabetes, active bleeding, ocular lesions Other serious diseases of the mental, nervous and other systems;
7. Clinically obvious digestive tract abnormalities during screening may affect drug intake, transport or absorption (such as dysphagia, uncontrollable nausea and vomiting, active gastric ulcers, ulcerative colitis, Crohn's disease, chronic diarrhea, intestinal obstruction, etc.);
8. Severe bone injury caused by tumor bone metastasis, with pathological fractures of important parts or spinal cord compression expected to occur in the near future within 6 months prior to knowledge;
9. There is cancerous meningitis or untreated central nervous system metastasis. Those who have previously received systemic or radical treatment for brain metastases (radiotherapy or surgery), and whose stability has been maintained for at least one month as confirmed by imaging, and who have stopped systemic hormone therapy (with a dose greater than 10mg/ day prednisone or other equivalent dose hormones) for more than two weeks and have no clinical symptoms, can be included;

9. There is cancerous meningitis or untreated central nervous system metastasis. Those who have previously received systemic or radical treatment for brain metastases (radiotherapy or surgery), and whose stability has been maintained for at least one month as confirmed by imaging, and who have stopped systemic hormone therapy (with a dose greater than 10mg/ day prednisone or other equivalent dose hormones) for more than two weeks and have no clinical symptoms, can be included 10.Patients with clinically symptomatic third space effusion (such as pleural effusion, ascites, pericardial effusion) who require puncture and drainage, or those who have received puncture and drainage within 2 weeks before the first medication; 11. At the time of screening, the toxicity of previous treatments had not yet recovered. According to CTCAE v5.0, there were still grade ≥2 AES (excluding special toxicities such as alopecia, fatigue, increased GGT, and increased ALP).

12. Have serious cardiovascular diseases, including but not limited to:

1. At rest, the 12-lead electrocardiogram examination showed that the QTcF was ≥470ms.
2. There are severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II-III degree atrioventricular block, etc.
3. Acute coronary syndrome, congestive heart failure (New York Heart Association (NYHA)) cardiac function grade ≥2, aortic dissection or other grade 3 cardiovascular events occurred within 6 months before the first administration.
4. Left ventricular ejection fraction (LVEF) <50%; 13. There is a history of thromboembolism or cerebrovascular events within 6 months before the first administration, including transient ischemic attack, cerebrovascular accident, deep vein thrombosis or pulmonary embolism, etc; 14. There was evidence of radiation pneumonitis, interstitial lung disease or interstitial pneumonia (ILD) requiring hormone therapy during the screening period, or drug-induced ILD, or any active ILD (such as acute exacerbation or progressive pneumonia/pulmonary fibrosis at baseline). Or pulmonary symptoms that the researchers consider unsuitable for enrollment, or high-risk factors that make it unsuitable for enrollment due to the possibility of interstitial lung disease; 15.Severe infection occurred within 4 weeks before the first administration, including but not limited to bacteremia and severe pneumonia that require hospitalization; There was an active infection of CTCAE grade ≥2 that required systemic antibiotic treatment within 2 weeks before the first administration (except for local chronic infections or prophylactic antibiotic use that the investigator determined did not require treatment).

   16. Those with a history of active pulmonary tuberculosis infection within 6 months prior to the first administration; 17. People infected with active human immunodeficiency virus (HIV), syphilis, hepatitis C virus (HCV) or hepatitis B virus (HBV). Active HBV, HCV and HIV infections are defined as:

a.positive HBsAg and HBV DNA ≥500cps/ml/HBV DNA ≥1000u/ml; b.Anti-hcv antibody and HCV RNA positive; c.HIV antibody positive. 18. Known history of alcohol or drug abuse or dependence; Mental disorder; Or the researcher believes that there is a history of other serious systemic diseases or other reasons that make the participants unsuitable for this study (such as not meeting the most beneficial treatment for the subjects, subject compliance, etc.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience one or more adverse events (AEs) | From Baseline up to 28 days after the end of the treatment
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Dose Limiting Toxicity (DLT) | Up to approximately 28 days
  Numbers of participants experiencing AEs which are defined as DLTs classfied by CTCAE v5.0.
Maximum tolerated dose（MTD） | Within 28 days of the first dose
  To determine the maximum tolerated dose for combination-agent escalation.
Recommended Phase 2 Dose（RP2D） | Within 28 days of the last patient dosed in escalation stage
  The RP2D is defined as the dose level chosen for the dose expansion arms, based on safety, tolerability, efficacy collected during the dose escalation portion of the study
Progression-free survival (rPFS） | Up to approximately 21 months
  rPFS is defined as the time from randomization to occurrence of: radiological tumor progression using RECIST 1.1 as assessed by BICR; progression of bone lesions using PCWG criteria; or death due to any cause. Progression as per modified RECIST 1.1 is ≥20% increase in the sum of diameters of target lesions and progression of existing non-target lesions. Progression of bone lesions by PCWG criteria is the appearance of ≥2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and are persistent for ≥6 weeks.

SECONDARY OUTCOMES:
Prostate-specific antigen (PSA) response rate | Up to approximately 21 months
  The Prostate-specific Antigen (PSA) response rate is the percentage of participants who had PSA response defined as a reduction in the PSA level from baseline by ≥50%. The reduction in PSA level will be confirmed by an additional PSA evaluation performed ≥3 weeks from the original response per Prostate Cancer Working Group (PCWG) criteria.
Overall survival (OS) | Up to approximately 21 months
  OS is defined as the time from randomization to death due to any cause.
Duration of response (DOR) | Up to approximately 21 months
  DOR is defined as the time from first documented evidence of complete response (CR) or partial response (PR) per PCWG and RECIST 1.1 criteria until progressive disease (PD) or death. PD per RECIST 1.1 is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of a least 5 mm. PD per PCWG is the appearance of >2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and are persistent for >6 weeks.
Objective response rate (ORR) | Up to approximately 21 months
  The ORR is defined as the percentage of participants with complete response (CR: disappearance of all target lesions per Response Criteria in Solid Tumors version 1.1 (RECIST 1.1); and no evidence of disease (NED) on base scan per Prostate Cancer Working Group (PCWG) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1; and non-progressive disease, non-evaluable [NE], or NED on bone scan or CR with non-progressive disease or NE bone scan per PCWG).

CONTACTS AND LOCATIONS:
Overall Officials: Ji Zhu, Doctor of Medicine, Principal Investigator — Doctor of Medicine; Doctor of Medicine, Principal Investigator — Zhejiang Cancer Hospital, Hangzhou, zhejiang
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No